CLINICAL TRIAL: NCT04240951
Title: Validity of a Prototype Wearable Patch in Measuring Local Sweating Rate and Sweat Electrolyte Concentration During Exercise
Brief Title: Sweat Patch Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1714
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Sweat Analysis
Keywords: sweating rate; sweat electrolytes; sweat patch; wearable; epidermal; sweat electrolyte concentrations

STUDY DESIGN:
Intervention Model Description: Each subject subject serves as their own control at each testing session. The prototype patch and reference method are both worn during each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Study Session 1 (Other): Arm Type: Validation. Regional sweat collection with prototype vs. reference patch in the laboratory
  Interventions: Other: Sweat patch
- Study Session 2 (repeat of Study Session 1) (Other): Arm Type: Validation: Regional sweat collection with prototype vs. reference patch in the laboratory
  Interventions: Other: Sweat patch
- Study Session 3 (Other): Arm Type: Validation. Prototype patch vs. whole body sweat collection in the laboratory
  Interventions: Other: Sweat patch
- Study Session 4 (repeat of Study Session 3) (Other): Arm Type: Validation. Prototype patch vs. whole body sweat collection in the laboratory
  Interventions: Other: Sweat patch
- Study Session 5 (Other): Arm Type: Validation. Regional sweat collection with prototype vs. reference patch in the field
  Interventions: Other: Sweat patch
- Study Session 6 (repeat of Study Session 5) (Other): Arm Type: Validation. Regional sweat collection with prototype vs. reference patch in the field
  Interventions: Other: Sweat patch

INTERVENTIONS:
Other: Sweat patch — Flexible, epidermal, wearable skin patch to collect and analyze sweat

SUMMARY:
To determine the validity of a prototype patch in measuring sweating rate and sweat electrolyte concentration during moderate intensity exercise against well-established reference methods in a controlled laboratory and in field conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* Subject is 15-45 years
* Subject is moderately-trained (engages in moderate-intensity, intermittent, or steady-state exercise at least 4 days per week for at least 1 hour at a time)
* Subject is capable of moderate-intensity, intermittent exercise for 1-2 hours as assessed by recent training history
* If participating in Study Session 1, 2, 3, or 4, subject has a treadmill VO2max ≥ 42 ml/kg/min if male or ≥ 38 ml/kg/min if female, as measured during the screening at the GSSI laboratory
* If participating in Study Session 1, 2, 3, or 4, subject has a normal fasting blood glucose (70-110 mg/dl), as measured during the screening at the GSSI laboratory
* If participating in Study Session 1, 2, 3, or 4, subject has a normal resting blood pressure (< 140/90 mmHg), as measured during the screening at the GSSI laboratory
* If participating in Study Session 1, 2, 3, or 4, subject has a normal resting and graded exercise EKG, as measured during the screening at the GSSI laboratory
* If participating in Study Session 1, 2, 3, or 4, willing to be shaved at patch sites
* If participating in Study Session 3 or 4, willing to undergo a nude shower by an investigator of the same sex for collection of sweat electrolytes in the whole body wash procedure
* If participating in Study Session 5 or 6, subject is a trained team-sport athlete currently participating in training/competition at IMG Academy

Exclusion Criteria:

* Subject is pregnant (self-reported)
* Subject is a smoker
* Subject has a body weight that is lighter than 80 pounds
* Subject has a known or suspected obstructive disease of the gastrointestinal tract, such as diverticulitis or inflammatory bowel disease
* Subject has a history of problems with the gag reflex
* Subject has not had previous gastrointestinal surgery
* Subject has problems with swallowing
* Subject is planning to have an MRI scan during the time that the CorTemp™ Core Body Temperature Sensor is in the body
* Subject has slow movement of the gastrointestinal tract
* Subject has a cardiac pacemaker or other implanted electronic device
* Subject has asthma or other condition in which breathing can become difficult/labored during exercise (applies to Study Session 1-4 only)
* Subject is allergic to adhesives
* Subject is currently taking a medication or oral supplement that could interfere with study results
* Subject has a condition the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk
* Subject has been enrolled into a PepsiCo-sponsored study within the past six months
* Subject has been enrolled into a clinical trial at a laboratory or clinic other than PepsiCo within the past 30 days
* Subject is employed by, or has a parent, guardian or other immediate family member employed by, a company that manufactures any products that compete with any Gatorade products. If subject is unsure if a company would be considered a competitor to Gatorade they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 552 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Sweat chloride concentration | 1.5 hours in sessions 1-6
  Prototype vs. reference method (regional absorbent patch technique) during exercise

SECONDARY OUTCOMES:
Regional sweating rate | 1.5 hours in sessions 1-6
  Prototype vs. reference method (gravimetry using the regional absorbent patch technique) during exercise
Whole body sweating rate | 1.5 hours in sessions 1-6
  Prototype vs. reference method (changes in nude body mass corrected for fluid intake, urine output, respiratory water loss, and metabolic mass loss) during exercise
Whole body sweat chloride concentration | 1.5 hours in sessions 3-4
  Prototype vs. reference method (whole body washdown technique) during exercise
Whole body sweat sodium concentration | 1.5 hours in sessions 3-4
  Reference method only. Compare whole body sweat chloride concentration vs. whole body sweat sodium concentration during exercise
Self-ratings of perceived sweating vs. measured sweating rate | Prior to the start of exercise at sessions 1-6
  Multiple choice questionnaire vs. sweat patch analysis
Self-ratings of perceived sweat saltiness vs. sweat electrolyte concentrations | Prior to the start of exercise at sessions 1-6
  Multiple choice questionnaire vs. sweat patch analysis
History of exercise-associated muscle cramps | Prior to the start of exercise at sessions 1-6
  Multiple choice questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay B Baker, PhD, Principal Investigator — PepsiCo Global R&D, Gatorade Sports Science Institute (GSSI) PI for Barrington site; Khalil Lee, PhD, Principal Investigator — PepsiCo Global R&D, Gatorade Sports Science Institute (GSSI) PI for Bradenton site
Locations (2):
- United States (2):
  - Gatorade Sports Science Institute at IMG Academy, Bradenton, Florida
  - Gatorade Sports Science Institute (GSSI), Barrington, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] King MA, Brown SD, Barnes KA, De Chavez PJD, Baker LB. Regional and time course differences in sweat cortisol, glucose, and select cytokine concentrations during exercise. Eur J Appl Physiol. 2023 Aug;123(8):1727-1738. doi: 10.1007/s00421-023-05187-3. Epub 2023 Apr 2. PMID 37005963